CLINICAL TRIAL: NCT02734264
Title: Field Studies of Human Immunity to Amebiasis in Bangladesh: A Prospective Study of Children Ages 0-17 Years
Brief Title: Field Studies of Amebiasis in Bangladesh
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, William Petri, MD, Division Chief, Infectious Disease, University of Virginia
Other Study IDs: 7563
Record Dates: First submitted 2016-03-22; First posted 2016-04-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-04

CONDITIONS: Amebiasis; Cryptosporidium
MeSH Terms: conditions — Amebiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and feces
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study will be to investigate the incidence of both Amebiasis and cryptosporidiosis in Bangladeshi children and examine genetic variation in innate and adaptive immunity with respect to these infections. Novel diagnostics to these infections will also be investigated.

DETAILED DESCRIPTION:
Entamoeba histolytica infection results from ingestion of the cyst of Entamoeba histolytica from fecally-contaminated food or water. Local invasion results in amebic dysentery and metastasis to amebic liver abscess. The diagnosis of intestinal amebiasis is ideally made using an E. histolytica-specific stool antigen detection test or using real-time polymerase chain reaction (PCR). The two major clinical syndromes of amebiasis are amebic colitis and amebic liver abscess. Together they are estimated to result in 50 million cases of colitis and liver abscess and 100,000 deaths worldwide each year. In developing countries, colonization with E. histolytica has been observed in 5% or more of poor children. Patients with amebic colitis typically present with a several week history of gradual onset of abdominal pain and tenderness, diarrhea and bloody stools (dysentery). The pathological lesions in the colon include ulceration of the intestinal epithelium and invasion into the lamina propria by trophozoites. Inflammation, with infiltrating neutrophils and mononuclear lymphocytes is pronounced, but inflammatory cells near the amebae are killed with pyknotic nuclei characteristic of apoptotic death. Amebic liver abscess is a rare form of the disease that is almost exclusively limited to adult males.

Cryptosporidiosis in humans is caused primarily by two species, Cryptosporidium parvum and C. hominis. There are annually approximately 1.4 cases/100,000 in the United States reported to the Centers for Disease Control. Infection results from ingestion of fecally contaminated water or food containing the infectious oocyst form. Sporozoites are released from the oocyst in the small intestine and attach to the epithelial cell surface. Upon invasion of the epithelial cells the parasite undergoes both the sexual and asexual stages of the life cycle. Infection with C. parvum in a normal host leads to days to several weeks of non-bloody diarrhea.

In many people E. histolytica and Cryptosporidia infections resolve without symptoms. A major emphasis of this study will be to study the host, environment, and parasite factors controlling susceptibility to E. histolytica and Cryptosporidia infection and disease, to begin to answer the question of why all infections do not cause disease. At the same time, want to improve diagnostic techniques for these diseases.

This study will continue a cohort of 420 children (average age now 10.5 years) that the research team has been following since birth and measure the incidence of amebiasis and cryptosporidiosis prospectively. In addition, 500 live births will be enrolled into an existing cohort.

This work has several objectives. The first objective is to compare current "gold-standard" diagnostic techniques for these diseases with newer antigen detection and polymerase chain reaction techniques. The second objective is to delineate the protective role of innate and acquired immunity to E. histolytica. The investigators hypothesize that protective immunity is mediated both by innate immune responses initiated via Toll-like Receptor stimulation and acquired responses including mucosal immunoglobulin A (IgA) and systemic Interferon-γ. Acquired immune responses (peripheral blood mononuclear cell cytokine production and fecal IgA anti-cross reacting determinant) during amebic and cryptosporidial infection and disease will be determined in the children in the cohort. The third objective is to test for the association of genetic polymorphisms in innate and acquired immune genes with incidence of amebiasis. The investigators hypothesize that common genetic polymorphisms in genes of the innate and acquired immune system influence susceptibility to E. histolytica and Cryptosporidia infection or disease. The final objective is to test the role of human genetic polymorphisms and microbiome in protection from undernutrition. Genome wide scans and microbiome compositional analyses will be performed on children to determine if the nutritional status of the child correlates with these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Mirpur, Dhaka, Bangladesh

Exclusion Criteria:

* Mother under 65 years old

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn children in the Mirpur neighborhood of Dhaka, Bangladesh.
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2008-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Amebiasis and Cryptosporidium infection | Birth to 5 years

SECONDARY OUTCOMES:
Peripheral blood mononuclear cell Interleukin (IL)-1β stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-2 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-4 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-5 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-6 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-7 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-8 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-10 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-12(p70) stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-12(p40) stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-13 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell IL-17 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell interferon-γ stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell granulocyte-macrophage colony-stimulating factor stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell tumor necrosis factor-α stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell tumor necrosis factor-β stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell granulocyte-colony stimulating factor stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell macrophage inflammatory protein (MIP)-1 β stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell MIP-1 α stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell monocyte chemotactic protein-1 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell eotaxin stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell fibroblast growth factor basic stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell vascular endothelial growth factor stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell "regulated on activation, normal T expressed and secreted" (RANTES) stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell leptin stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell epithelial neutrophil activating peptide (ENA)-78 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell nerve growth factor stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Peripheral blood mononuclear cell inducible protein-10 stimulation studies | Birth to 5 years
  Investigators plan to obtain blood for cytokine analysis from children when they do not have E. histolytica infection and are free of diarrheal disease. Investigators also plan to obtain blood for cytokine analysis from children within 48 hours of the diagnosis of E. histolytica infection or disease.
Fecal immunoglobulin-A | Birth to 5 years
  This will be collected as paired samples. One sample will be from each episode of Amebiasis diarrhea and will paired with a stool from that child when they have no Amebiasis detected in the stool and are without acute diarrhea.
Fecal immunoglobulin-G anti-cross-reacting determinant | Birth to 5 years
  This will be collected as paired samples. One sample will be from each episode of Amebiasis diarrhea and will paired with a stool from that child when they have no Amebiasis detected in the stool and are without acute diarrhea.
Single nucleotide polymorphism analysis of innate and adaptive immunity | Once; between birth and day 7 of life.
Genome wide association scan | Once, at 5 years of age
Fecal microbiome determination via 16s ribosomal deoxyribonucleic acid (rDNA) | Birth to 5 years
Length/Height in centimeters | Birth to 5 years
Weight in grams | Birth to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William A Petri, M.D., PhD, Principal Investigator — University of Virginia
Locations (1):
- The International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Zhou J, Niu F, Donowitz JR, Haque R, Petri WA Jr, Ma JZ. Characterizing early child growth patterns of height-for-age in an urban slum cohort of Bangladesh with functional principal component analysis. BMC Pediatr. 2017 Mar 21;17(1):84. doi: 10.1186/s12887-017-0831-y. PMID 28327104